CLINICAL TRIAL: NCT01224249
Title: Selenium Status Measured in Blood After a Higher Intake of Fish and Shellfish - a Randomized Dietary Intervention Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Danish Cancer Society (Other)
Collaborators: Technical University of Denmark (Other); Danish Shellfish Center (Other)
Responsible Party: Anne Tjønneland, professor, M.D., Ph.D., Institute of Cancer Epidemiology, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DCS-53227244
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-08

CONDITIONS: Selenium Status; Selenium Uptake From Fish and Shellfish
Keywords: Selenium; Selenoprotein P; Fish; Shellfish; Bioavailability
MeSH Terms: interventions — In Situ Hybridization, Fluorescence; Shellfish

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish and shellfish (Active Comparator)
  Interventions: Dietary Supplement: Fish and shellfish
- Control (No Intervention): Assessment only

INTERVENTIONS:
Dietary Supplement: Fish and shellfish — Intake of 1000 grams of fish and shellfish per week for six months.
  Arms: Fish and shellfish

SUMMARY:
The primary aim of this study is to investigate, whether higher intake of selenium rich food items such as fish and shellfish, is associated with higher selenium blood levels.

The secondary aim is to investigate the uptake of selenium from fish and shellfish and the incorporation of selenium from those foods into proteins in the human body. Furthermore, the impact of the natural variation in the genes that are responsible for the accumulation of selenium in the proteins will be investigated.

DETAILED DESCRIPTION:
Selenium is an essential trace element that is incorporated into proteins in the human body and it hereby plays a major role in several important cellular processes. Previous studies have indicated that the selenium status of the Danish population is below the levels required to optimize the suggested protective effects of selenium towards major diseases including cancer. In Denmark, important natural sources of selenium are fish and shellfish.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* 50-74 years
* BMI 18.5-28 kg/m2
* non-smokers

Exclusion Criteria:

* strenuous exercise > 10 h/week
* excessive intake of alcohol
* frequent intake of fish and shellfish > 200-300 g/week
* intake of dietary supplements 3 months before or during the study
* frequent use of medication except antihypertensive medicine, cholesterol lowering medicine and hormone replacement medicine
* simultaneous participation in other research projects
* cancer diagnosis within the past 5 years
* severe chronic diseases

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Selenium concentration in whole blood | Measured at baseline
Selenium concentration in whole blood | Measured after 3 months of intervention
Selenium concentration in whole blood | Measured after 6 months of intervention

SECONDARY OUTCOMES:
Selenoprotein P in plasma | Measured at baseline
Selenoprotein P in plasma | Measured after 3 months of intervention
Selenoprotein P in plasma | Measured after 6 months of intervention
Genetic polymorphisms in the selenoprotein P gene | Measured at baseline
Genetic polymorphisms in the selenoprotein P gene | Measured after 3 months of intervention
Genetic polymorphisms in the selenoprotein P gene | Measured after 6 months of intervention
Heavy metals in whole blood (lead, cadmium, and mercury) | Measured at baseline
Heavy metals in whole blood (lead, cadmium, and mercury) | Measured after 3 months of intervention
Heavy metals in whole blood (lead, cadmium, and mercury) | Measured after 6 months of intervention
Blood pressure | Measured at baseline
Blood pressure | Measured after 3 months of intervention
Blood pressure | Measured after 6 months of intervention
Anthropometry (weight, height, waist, and hip circumference) | Measured at baseline
Anthropometry (weight, height, waist, and hip circumference) | Measured after 3 months of intervention
Anthropometry (weight, height, waist, and hip circumference) | Measured after 6 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anne Tjonneland, professor, M.D., Ph.D., Principal Investigator — Institute of Cancer Epidemiology, Danish Cancer Society
Locations (1):
- Institute of Cancer Epidemiology, Danish Cancer Society, Copenhagen, Denmark